CLINICAL TRIAL: NCT03491020
Title: Emission Patterns of Respiratory Pathogens
Status: Withdrawn | Type: Observational
Why Stopped: Trial has been withdrawn due to logistical support issues.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00038054
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-06

CONDITIONS: Pathogen Transmission
Keywords: Emission Patterns; Respiratory; Aerosolization; Airborne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The results of routine in-house laboratory diagnostic tests such as the Respiratory Viral Panel (RVP), serology tests or bacterial cultures will be used to identify patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Respiratory syncytial virus (RSV): Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify RSV.
- Enteroviruses: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify enterovirus.
- Adenoviruses: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify adenovirus.
- Coronaviruses: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify coronavirus.
- Metapneumoviruses: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify metapneumovirus.
- Chlamydia pneumoniae: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify chlamydia pneumoniae.
- Mycoplasma: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify mycoplasma.
- Parainfluenza: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify parainfluenza.
- Neisseria meningitides: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify neisseria meningitides.
- Bordetella pertussis: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify bordetella pertussis.
- Rhinovirus: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with a respiratory pathogen. A nasopharyngeal swab will be obtained to identify rhinovirus.

SUMMARY:
Airborne transmission represents one of the most rapidly spreading and dangerous dissemination mechanisms for pathogens. Public health strategies to prevent and control the often explosive outbreaks associated with such pathogens are: 1) vaccination and treatment, if available, 2) isolation and barrier precautions such as face masks, and 3) decontamination of the exposed areas and surfaces. A lack of understanding how these pathogens are transmitted hampers the ability to develop effective prevention measures. This study will be used to collect preliminary data of the emission patterns of respiratory pathogens.

DETAILED DESCRIPTION:
Airborne transmission represents one of the most rapidly spreading and dangerous dissemination mechanisms for pathogens. The study team have been investigating bacterial and viral transmission routes and barrier precautions. In a recent clinical study, it was observed that Measles virus RNA was detected from a patient for at least up to 10 feet. In addition, the group has been studying barrier precautions (facemasks) for their ability to prevent the spread of aerosolized viruses. Finally, in a controlled lab setting the investigators have assessed the impact of environmental conditions (temperature, humidity) on pathogen transmission and the effect of UV-C light to prevent the spread of influenza. The purpose of this observational study is to describe the human aerosolization patterns of respiratory pathogens. The study team hypothesizes that the emission patterns of specific airborne pathogens varies between individual patients.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years of age admitted to the ED or an inpatient care unit of Wake Forest Baptist Medical Center (WFBMC)
* Positive

Exclusion Criteria:

* positive respiratory pathogen tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years of age admitted to the ED or an inpatient care unit of Wake Forest Baptist Medical Center (WFBMC) will be screened for respiratory pathogens (performed as part of standard clinical care). Participants with positive respiratory pathogen tests will be consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
particle size distribution patterns: ICU | throughout study completion, up to 7 days
  This outcome measure will determine the particle size distribution patterns of the pathogen in the intensive care unit (ICU).
particle size distribution patterns: non-ICU setting | throughout study completion, up to 7 days
  This outcome measure will determine the particle size distribution patterns of the pathogen in the non-intensive care unit (ICU).
quantities of the pathogen: ICU | throughout study completion, up to 7 days
  This outcome measure will determine the quantities of the pathogen in the intensive care unit (ICU).
quantities of the pathogen: non-ICU setting | throughout study completion, up to 7 days
  This outcome measure will determine the quantities of the pathogen in the non-intensive care unit (ICU).
spatial model: ICU | throughout study completion, up to 7 days
  This outcome measure will establish a spatial model (1 foot vs. 3- feet vs. 8-10 feet) of airborne pathogen dispersal in the ICU.
spatial model: non-ICU setting | throughout study completion, up to 7 days
  This outcome measure will establish a spatial model (1 foot vs. 3- feet vs. 8-10 feet) of airborne pathogen dispersal in a non-ICU setting.
correlation between the human aerosolization patterns and the severity of illness | throughout study completion, up to 7 days
  This outcome measure is to determine the correlation between the human aerosolization patterns and the severity of illness (fever, respiratory symptoms, malaise) in individual participants.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Bischoff, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.